CLINICAL TRIAL: NCT01369836
Title: An Investigator And Subject-Blind Phase 1 Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-06291826 (Tafamidis) After Single Oral Administration To Japanese And Western Healthy Subjects
Brief Title: Study Of Single Doses Of PF-06291826 (Tafamidis) In Japanese And Western Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B3461009
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Tafamidis; Pharmacokinetics; TTR stabilization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg soft gelatin capsule (Experimental)
  Interventions: Drug: Tafamidis meglumin
- 40 mg (20 mg*2) soft gelatin capsule (Experimental)
  Interventions: Drug: Tafamidis meglumin
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafamidis meglumin — A single oral dose of 20 mg capsule
  Other Names: PF-06291826
  Arms: 20 mg soft gelatin capsule
Drug: Tafamidis meglumin — A single oral dose of 40 mg capsule.
  Other Names: PF-06291826
  Arms: 40 mg (20 mg*2) soft gelatin capsule
Drug: Placebo — A single oral dose of matched placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is the following:

* To evaluate the safety, tolerability, and pharmacokinetics (PK) of orally administered tafamidis in Japanese and Western healthy volunteers at single dose.
* To compare Japanese and Western PK profiles.
* Determine the PD stabilization effect of tafamidis on human transthyretin (TTR) in a validated ex vivo assay.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.

Exclusion Criteria:

* Pregnant or nursing females.
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of tafamidis over time (AUClast). | 2 months
Plasma concentration of tafamidis over time (Cmax). | 2 months
Plasma concentration of tafamidis over time (Tmax). | 2 months
If data permit, AUCinf and t1/2 will be determined. | 2 months

SECONDARY OUTCOMES:
The percent stabilization of TTR tetramer will be defined at Cmax in each subject and compared between Japanese volunteers and Western volunteers. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461009&StudyName=Study%20Of%20Single%20Doses%20Of%20PF-06291826%20%28Tafamidis%29%20In%20Japanese%20And%20Western%20Subjects